CLINICAL TRIAL: NCT03018197
Title: The Use of Electronic Personal Health Records to Improve Medication Adherence Among Non-Valvular Atrial Fibrillation Patients: A Pilot Study
Brief Title: Use of Electronic Personal Health Records to Improve Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkview Health (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Mirro, Chief Academic and Research Officer, Parkview Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRC13-0806 ePHR AFib pilot
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation; Medication Adherence
Keywords: Personal Health Record; Medication Knowledge; Anticoagulants; Patient Engagement
MeSH Terms: conditions — Atrial Fibrillation; Medication Adherence; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medication Education (Experimental): Patients will receive training on the use of the personal health record and health education via the personal health record.
  Interventions: Other: Medication Education
- No Medication Education (No Intervention): Patients will receive the current standard of care for the personal health record. Patients will not receive training on the use of the personal health record or health education via the personal health record.

INTERVENTIONS:
Other: Medication Education — Medication education delivered via the personal health record (MyChart) pertinent to the anticoagulation medication dabigatran. Education newsletters will be sent at 4, 6, and 10 weeks post-enrollment.
  Arms: Medication Education

SUMMARY:
The purpose of this pilot study is to examine the use of a personal health record to improve medication adherence among patients with non-valvular atrial fibrillation taking dabigatran for primary prevention of embolic stroke.

DETAILED DESCRIPTION:
Three brief newsletters will be sent by the research staff to the study patients in the form of secure messages through their MyChart account. The newsletters will describe dabigatran tolerability, adverse effects, patient monitoring, warnings/precautions, and administration. Newsletters will be developed through a review of the FDA-approved prescribing information, general tertiary references, and a search of PubMed and drafted with guidance from a Drug Information Specialist at Manchester University College of Pharmacy as well as reviewed by the research staff.

Descriptive analysis will be used to analyze the survey to assess patient attitudes and beliefs about dabigatran and personal health records, as well as to assess the level of patient engagement. Difference-in-difference regression analysis will be used to evaluate the impact of the personal health record on dabigatran adherence by comparing the differences between times (pre-post) and interventions. Patient medication adherence will be correlated from the Pharmacy refill data to determine if the Intervention Group is more compliant than the Control Group. Multivariate analysis will be used to explore factors influencing personal health record use and dabigatran adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient of Parkview Physicians Group-Cardiology
* Currently on dabigatran for non-valvular atrial fibrillation
* Out-patient status
* Ability to read and understand English
* Access to the Internet
* Ability to utilize the computer and Internet
* Willingness to enroll in a MyChart account

Exclusion Criteria:

* Physical or cognitive disability hindering provision of the informed consent process or performance of study tasks
* Unable to physically or cognitively carry out the tasks necessary for activating and/or utilizing a personal health record
* Designated as part of a vulnerable subject population that the investigator or designee identifies to have compromised autonomy related to potential study participation
* Currently part of another study involving another type of personal health record (other than MyChart)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Medication Adherence evaluated through medication possession ratios | 3 months during study

SECONDARY OUTCOMES:
Patient Engagement evaluated through Patient Activation Measure (PAM) | 3 months during study
Medication Knowledge evaluated through 5-question survey | 3 months during study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mirro, MD, Principal Investigator — Parkview Health; Ozlem Ersin, PhD, Principal Investigator — Manchester University College of Medicine
Locations (1):
- Parkview Research Center; Parkview Health, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.